CLINICAL TRIAL: NCT06066528
Title: A Phase 3, Randomised, Double-blind, Parallel-group, 76-week, Efficacy and Safety Study of BI 456906 Administered Subcutaneously Compared With Placebo in Participants With Overweight or Obesity and Type 2 Diabetes Mellitus
Brief Title: A Study to Test Whether Survodutide (BI 456906) Helps People Living With Overweight or Obesity Who Also Have Diabetes to Lose Weight
Acronym: SYNCHRONIZE™-2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1404-0041; 2022-502531-18-00 (Registry Identifier: CTIS); U1111-1289-0247 (Registry Identifier: WHO registry)
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Obesity; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — BI 456906

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Survodutide 3.6 mg (Experimental)
  Interventions: Drug: Survodutide
- Survodutide 6.0 mg (Experimental)
  Interventions: Drug: Survodutide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Survodutide — once weekly subcutaneous injection
  Other Names: BI 456906
  Arms: Survodutide 3.6 mg; Survodutide 6.0 mg
Drug: Placebo — once weekly subcutaneous injection
  Arms: Placebo

SUMMARY:
This study is open to adults who are at least 18 years old and have a body mass index of 27 kg/m² or more. People can take part if they have type 2 diabetes and if they are currently being treated only with diet and exercise or with specific diabetes medications. Only people who have previously not managed to lose weight by changing their diet can participate.

The purpose of this study is to find out whether a medicine called survodutide (BI 456906) helps people living with overweight or obesity who also have diabetes to lose weight.

Participants are divided into 3 groups by chance, like drawing names from a hat. 2 groups get different doses of survodutide and 1 group gets placebo. Placebo looks like survodutide but does not contain any medicine. Every participant has a 2 in 3 chance of getting survodutide. Participants inject survodutide or placebo under their skin once a week for about one and a half years. In addition to the study medicine, all participants receive counselling to make changes to their diet and to exercise regularly.

Participants are in the study for about 1 year and 7 months. During this time, it is planned that participants visit the study site up to 14 times and receive 6 phone calls by the site staff.

The doctors check participants' health and take note of any unwanted effects. The study staff also regularly measure participants' body weight. The results are compared between the groups to see whether the treatment works.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥18 years at the time of signing informed consent, and at least the legal age of consent in countries where it is >18 years.
2. Body mass index (BMI) ≥27 kg/m^2 at screening.
3. Diagnosed with Type 2 diabetes mellitus (T2DM) (defined as Glycosylated haemoglobin A1c (HbA1c) ≥6.5% [≥48 mmol/mol]) at least 180 days prior to screening.
4. HbA1c ≥6.5% (≥48 mmol/mol) and <10% (<86 mmol/mol) as measured by the central laboratory at screening.
5. Currently treated for T2DM with either diet and exercise alone or stable treatment (for at least 3 months prior to screening) per treatment guidelines.
6. History of at least one self-reported unsuccessful dietary effort to lose body weight Further inclusion criteria apply.

Exclusion Criteria:

1. Body weight change (self-reported) of >5% within 3 months before screening.
2. Treatment with any medication for the indication obesity within 3 months before screening.
3. Treatment with any medication for indication of T2DM other than stated in the inclusion criteria and glucagon-like peptide-1 receptor (GLP-1R)-based agonists) and dipeptidyl peptidase 4 inhibitor [DPP-4il).
4. Known clinically significant gastric emptying abnormality (e.g., severe diabetic gastroparesis or gastric outlet obstruction).
5. History of either chronic or acute pancreatitis or elevation of serum lipase or amylase >2x upper limit of normal (ULN)) as measured by the central laboratory at screening.
6. Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN 2).

Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 755 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2026-04-03 (Estimated)

PRIMARY OUTCOMES:
Percentage change in body weight from baseline to Week 76 | Baseline and at Week 76
Achievement of body weight reduction ≥5% (yes/no) from baseline to Week 76 | Baseline and at Week 76

SECONDARY OUTCOMES:
Achievement of body weight reduction ≥10% (yes/no) from baseline to Week 76 | Baseline and at Week 76
Achievement of body weight reduction ≥15% (yes/no) from baseline to Week 76 | Baseline and at Week 76
Achievement of body weight reduction ≥20% (yes/no) from baseline to Week 76 | Baseline and at Week 76
Absolute change from baseline to Week 76 in body weight (kg) | Baseline and at Week 76
Absolute change from baseline to Week 76 in glycosylated haemoglobin A1c (HbA1c) (%) | Baseline and at Week 76
Absolute change from baseline to Week 76 in waist circumference (cm) | Baseline and at Week 76
Absolute change from baseline to Week 76 in systolic blood pressure (SBP) (mmHg) | Baseline and at Week 76
Absolute change from baseline to Week 76 in "Capacity to Resist" domain score of Eating Behaviour patient reported outcome (PRO) | Baseline and at Week 76
  "Capacity to Resist" domain score of the Eating Behaviour PRO is ranging between 0 and 24 and a higher score indicates a lower capacity to resist.
Key secondary endpoint: Absolute change from baseline to Week 76 in Eating Behaviour PRO total score | Baseline and at Week 76
  Eating Behaviour PRO total score is ranging between 0 and 48 and a higher score indicates a worse eating behaviour (greater desire to eat and/or lower capacity to resist).
Absolute change from baseline to Week 76 in body mass index (BMI) (kg/m2) | Baseline and at Week 76
Absolute change from baseline to Week 76 in HbA1c (mmol/mol) | Baseline and at Week 76
Absolute change from baseline to Week 76 in diastolic blood pressure (DBP) (mmHg) | Baseline and at Week 76
Absolute change from baseline to Week 76 in fasting plasma glucose (FPG) (mg/dL) | Baseline and at Week 76
Absolute change from baseline to Week 76 in fasting plasma insulin (FPI) (mIU/L) | Baseline and at Week 76
Absolute change from baseline to Week 76 in total cholesterol (mg/dL) | Baseline and at Week 76
Absolute change from baseline to Week 76 in high density lipoprotein (HDL) cholesterol (mg/dL) | Baseline and at Week 76
Absolute change from baseline to Week 76 in low density lipoprotein (LDL) cholesterol (mg/dL) | Baseline and at Week 76
Absolute change from baseline to Week 76 in very-low-density lipoprotein (VLDL) cholesterol (mg/dL) | Baseline and at Week 76
Absolute change from baseline to Week 76 in triglycerides (mg/dL) | Baseline and at Week 76
Absolute change from baseline to Week 76 in free fatty acids (mg/dL) | Baseline and at Week 76
Absolute change from baseline to Week 76 in alanine aminotransferase (ALT) (U/L) | Baseline and at Week 76
Absolute change from baseline to Week 76 in aspartate aminotransferase (AST) (U/L) | Baseline and at Week 76

CONTACTS AND LOCATIONS:
Locations (143):
- United States (34):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - EmVenio Research-Atlanta-69582, Phoenix, Arizona
  - Encompass Clinical Research, Spring Valley, Spring Valley, California
  - Diablo Clinical Research, Walnut Creek, California
  - Alliance for Multispecialty Research, LLC - Doral, Doral, Florida
  - University of Florida, Gainesville, Florida
  - East Coast Institute for Research, LLC - Jacksonville, Jacksonville, Florida
  - New Horizon Research Center-Miami-69732, Miami, Florida
  - West Orange Endocrinology, Ocoee, Florida
  - Emory University, Atlanta, Georgia
  - East-West Medical Research, Honolulu, Hawaii
  - Solaris Clinical Research, Meridian, Idaho
  - Evanston Premier Healthcare Research LLC, Skokie, Illinois
  - Velocity Clinical Research-Valparaiso-68883, Valparaiso, Indiana
  - Velocity Clinical Research-Sioux City-69728, Sioux City, Iowa
  - AMR Lexington, Lexington, Kentucky
  - L-MARC Research Center, Louisville, Kentucky
  - StudyMetrix Research, LLC, City of Saint Peters, Missouri
  - Walgreens Clinical Trials-Atlantic City-69647, Atlantic City, New Jersey
  - Walgreens - Perth Amboy - Site 4544, Perth Amboy, New Jersey
  - Premier Research, Inc., Trenton, New Jersey
  - Velocity Clinical Research - Binghamton, Binghamton, New York
  - Southgate Medical Group/ Southgate Medical Park, West Seneca, New York
  - Physicians East, PA, Greenville, North Carolina
  - Lucas Research, Inc., Morehead City, North Carolina
  - Accellacare-Wilmington-67123, Wilmington, North Carolina
  - EmVenio Research-Oklahoma City-70053, Oklahoma City, Oklahoma
  - Trial Management Associates, Myrtle Beach, South Carolina
  - Texas Diabetes and Endocrinology, Austin, Texas
  - Juno Research, LLC, Houston, Texas
  - Diabetes & Glandular Disease Clinic, P.A., San Antonio, Texas
  - Consano Clinical Research, Shavano Park, Texas
  - Manassas Clinical Research Center, Manassas, Virginia
  - Rainier Clinical Research Center, Renton, Washington
- Australia (8):
  - Nepean Hospital, Kingswood, New South Wales
  - Hunter Diabetes Centre, Merewether, New South Wales
  - CORE Research Group, Milton, Queensland
  - Griffith Health, Southport, Queensland
  - Monash University, Box Hill, Victoria
  - Austin Health, Heidelberg, Victoria
  - Baker Heart and Diabetes Institute, Melbourne, Victoria
  - Keogh Institute for Medical Research, Nedlands, Western Australia
- Belgium (3):
  - ASZ - Campus Aalst, Aalst
  - UZ Leuven, Leuven
  - Roeselare - HOSP AZ Delta, Roeselare
- Canada (11):
  - Centricity Research (Calgary), Calgary, Alberta
  - Dr. James Lai, Vancouver, British Columbia
  - Aggarwal and Associates Ltd., Brampton, Ontario
  - The Wharton Medical Clinic Clinical Trials Inc., Hamilton, Ontario
  - Milestone Research Inc., London, Ontario
  - James Cha, MD, Oshawa, Ontario
  - Stouffville Medical Research Institute Inc., Stouffville, Ontario
  - Albion Finch Medical Centre, Toronto, Ontario
  - Sameh Fikry Medicine Professional Corporation, Waterloo, Ontario
  - Recherche GCP Research, Montreal, Quebec
  - Power Clinical Research, Montreal, Quebec
- China (20):
  - Peking University People's Hospital, Beijing
  - Beijing Pinggu Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Changzhou Second People's Hospital, Changzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - Forth Clinical Hospital of Harbin Medical University, Harbin
  - Huzhou Central Hospital, Huzhou
  - Center Hospital of Jinan, Jinan
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing
  - Pingxiang People's Hospital, Pingxiang
  - Shanghai Municipal Hospital of Traditional Chinese Medicine, Shanghai
  - Shanghai Fifth People's Hospital affiliated to Fudan University, Shanghai
  - Siping Central People's Hospital, Siping
  - Suzhou Municipal Hospital, Suzhou
  - Tianjin Medical University General Hospital, Tianjin
  - Wuhan Union Hospital, Wuhan
  - The First Affiliated Hospital of Xi'an Medical University, Xi'an
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Affiliated Hospital of Jiangsu University, Zhenjiang
- Czechia (5):
  - EDUMED s.r.o., Náchod
  - NZZ Agentura Science Pro s.r.o., Olomouc, Olomouc
  - Dieko, s.r.o., Pilsen
  - Polyclinic Michnova Ltd., Prague
  - Private Practice - Dr. Barbora Diepoltova, Prague
- Sanos Clinic Gandrup (SMO), Gandrup, Denmark
- Finland (3):
  - HUS, Lihavuustutkimusyksikkö Biomedicum Helsinki, Helsinki
  - Itä-Suomen yliopisto/Health Step Finland Oy, Kuopio
  - CRST - Clinical Research Services Turku, Turku
- Germany (6):
  - InnoDiab Forschung GmbH, Essen
  - MVZ im Altstadt-Caree Fulda GmbH, Fulda
  - Diabetes Zentrum Hamburg West, Hamburg
  - Institut für Diabetesforschung Münster GmbH, Münster
  - R.E.D. Institut fuer medizinische Studien und Fortbildung GmbH, Oldenburg in Holstein
  - Forschungszentrum Ruhr, KliFo Center GmbH, Witten
- Greece (3):
  - Athens Medical Center, Athens
  - Thermi Clinic, Thermi
  - Nexthealth S.A, Thessaloniki
- Hungary (5):
  - DRC Drug Research Ltd-Balatonfured-59734, Balatonfüred
  - Belinus Bt, Debrecen
  - CRU Hungary Ltd., Kistarcsa
  - Arina Trial Research kft., Orosháza
  - University of Szeged, Szeged
- Japan (6):
  - Fukuhama Chuo Clinic, Fukuoka, Fukuoka
  - Itabashi Diabetic medicine and Dermatology Clinic, Ibaraki, Koga
  - Noritake Clinic, Ibaraki, Ushiku
  - Soka Sugiura Naika Clinic, Saitama, Soka
  - Oyama East Clinic, Tochigi, Oyama
  - Hachioji Diabetes Clinic, Tokyo, Hachioji
- Netherlands (2):
  - PT & R, Born
  - Universitair Medisch Centrum Groningen, Groningen
- New Zealand (5):
  - P3 Research Dunedin, Dunedin
  - Southern Clinical Trials Tasman, Nelson
  - P3 Research-Newtown Wellington NZ-33770, Newtown Wellington NZ
  - Optimal Clinical Trials North, Rosedale, Auckland
  - P3 Research-Tauranga-34833, Tauranga
- Poland (5):
  - PI HOUSE Sp. z o.o., Gdansk, Gdansk
  - ETG Lublin, Lublin
  - Velocity Nova Sp z o.o., Puławy
  - ETG Siedlce, Siedlce
  - Clinical Research Center METABOLICA lek. Robert Witek, Tarnów
- South Korea (9):
  - The Catholic University of Korea, Bucheon St.Mary's Hospital, Bucheon-si
  - Kyungpook National University Hospital, Daegu
  - Dongguk University Ilsan Hospital, Goyang
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - The Catholic University of Korea, Yeouido St.Mary's Hospital, Seoul
  - Ajou University Hospital, Suwon
- Spain (7):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Vithas Sevilla, Castilleja de la Cuesta
  - Hospital Arnau de Vilanova, Lleida
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Clínica Universidad de Navarra - Madrid, Madrid
  - Clínica Universidad de Navarra, Pamplona
  - Hospital de Canarias, San Cristóbal de La Laguna
- Sweden (5):
  - Ladulaas Kliniska Studier, Borås
  - Forskningsenheten Carlanderska, Gothenburg
  - Pharmasite Malmo, Malmo
  - Medicinmottagning 5/Överviktsenheten, Örebro
  - Sabbatsbergs sjukhus, Stockholm
- United Kingdom (5):
  - Waterloo Medical Centre, Blackpool
  - Bradford on Avon Health Centre, Bradford-on-Avon
  - Mounts Bay Medical Limited, Hayle
  - Clifton Medical Centre, Rotherham, Rotherham
  - Trowbridge Health Centre, Trowbridge

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section 'time frame' are fulfilled, researchers can use the following link https:// www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After structured results have been posted, all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'.For study data -1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing

REFERENCES:
- [Derived] Wharton S, le Roux CW, Bozkurt B, Platz E, Bleckert G, Ajaz Hussain S, Brueckmann M, Startseva E, Kloer IM, Kaplan LM. Baseline characteristics in the SYNCHRONIZE-2 randomized phase 3 trial of survodutide, a glucagon receptor/GLP-1 receptor dual agonist, for obesity in people with type 2 diabetes. Diabetes Obes Metab. 2026 Feb;28(2):1490-1498. doi: 10.1111/dom.70263. Epub 2025 Nov 11. PMID 41216778
- See also: Related Info — http://www.mystudywindow.com